CLINICAL TRIAL: NCT07280533
Title: Accuracy of Virtual Surgical Planning in Reduction of Zygomatico-Maxillary Fractures A Randomized Clinical Controlled Study
Brief Title: Accuracy of Virtual Surgical Planning Versus Traditional Technique in Zygomaticomaxillary Fracture Reduction
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Suez Canal University (Other)
Collaborators: Suez canal university hospitals (Unknown)
Responsible Party: Principal Investigator, hossam shaban, Principal Investigator, Department of Oral and Maxillofacial Surgery, Suez Canal University, Suez Canal University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1002/2025
Record Dates: First submitted 2025-11-14; First posted 2025-12-12 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Facial Bone Fracture; Maxillofacial Injury; Zygomaticomaxillary Complex Fracture
Keywords: Zygomaticomaxillary complex fracture; ZMC fracture; Virtual surgical planning; 3D printing; Prebent titanium miniplates; Facial symmetry; Computer-assisted surgery; CT evaluation; Traditional surgical method
MeSH Terms: conditions — Maxillofacial Injuries | interventions — Fracture Fixation, Internal

STUDY DESIGN:
Intervention Model Description: clinical trial compares two different surgical approaches for treating zygomaticomaxillary complex (ZMC) fractures):
  Experimental Arm (Group I):
  Virtual surgical planning (VSP) with 3D model printing and prebent titanium miniplates.
  Active Comparator Arm (Group II):
  Traditional open reduction and fixation without virtual planning or prebent plates.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Surgical Planning (VSP) - Prebent Miniplates (Experimental): Patients allocated to this arm will undergo preoperative CT segmentation and 3D reconstruction, virtual reduction of the zygomaticomaxillary complex, and 3D printing of the reduced model. Titanium miniplates will be prebent on the 3D printed model before surgery. Surgical fixation will then be performed under general anesthesia using the prebent titanium miniplates.
  Interventions: Procedure: Virtual surgical planning and 3D model printing; Device: Prebent titanium miniplates
- Traditional Open Reduction and Fixation (Active Comparator): Patients allocated to this arm will undergo conventional open reduction and internal fixation of the ZMC fracture under general anesthesia without prior virtual surgical planning or 3D-printed models. Titanium miniplates will be contoured intraoperatively by the surgical team and used for fixation at the appropriate sites.
  Interventions: Procedure: Conventional open reduction and internal fixation (ORIF); Device: Titanium miniplates and screws (Anton Hipp)

INTERVENTIONS:
Procedure: Virtual surgical planning and 3D model printing — Preoperative CT segmentation, virtual reduction of fracture fragments using 3D planning software, and printing of the reduced 3D anatomical model for plate prebending.
  Arms: Virtual Surgical Planning (VSP) - Prebent Miniplates
Device: Prebent titanium miniplates — Titanium miniplates prebent on the printed model and used for rigid internal fixation at standard zygomatic fixation points (frontozygomatic suture, infraorbital rim, zygomaticomaxillary buttress) as indicated.
  Arms: Virtual Surgical Planning (VSP) - Prebent Miniplates
Procedure: Conventional open reduction and internal fixation (ORIF) — Standard surgical exposure and manual reduction of fracture fragments with intraoperative confirmation of alignment, followed by contouring and application of titanium miniplates and screws for fixation.
  Arms: Traditional Open Reduction and Fixation
Device: Titanium miniplates and screws (Anton Hipp) — Surgeon-contoured titanium miniplates applied intraoperatively at the necessary fixation points.
  Arms: Traditional Open Reduction and Fixation

SUMMARY:
This randomized clinical trial aims to evaluate the accuracy and outcomes of virtual surgical planning (VSP) compared to the traditional surgical technique in the reduction of zygomaticomaxillary complex (ZMC) fractures. Twenty patients with ZMC fractures will be randomly assigned into two equal groups: one treated using virtual planning and prebent titanium miniplates, and the other treated conventionally without virtual planning. Clinical evaluation will include facial symmetry, eye movement, and postoperative complications, while radiographic assessment will be performed using CT scans three months after surgery to measure bone formation and alignment accuracy. The study seeks to determine whether virtual surgical planning improves anatomical restoration, esthetics, and functional outcomes compared to traditional methods.

DETAILED DESCRIPTION:
Background:

The zygomaticomaxillary complex (ZMC) is one of the most frequently fractured regions of the facial skeleton due to its prominent anatomical position. Improper reduction can lead to functional impairment, facial asymmetry, and poor esthetic results. Virtual surgical planning (VSP) and 3D printing have recently been introduced to enhance surgical precision through preoperative simulation and prebending of fixation plates. However, the clinical superiority of this technique over traditional surgical methods remains under investigation.

Objective:

To compare the accuracy and clinical outcomes of virtual surgical planning and prebent titanium miniplates versus conventional open reduction and internal fixation techniques in the management of zygomaticomaxillary complex fractures.

Methods:

This randomized clinical trial will include 20 patients diagnosed with unilateral ZMC fractures, divided equally into two groups.

Group I: Patients treated using virtual surgical planning with 3D model reconstruction, virtual reduction, and prebending of titanium miniplates.

Group II: Patients treated using traditional open reduction and fixation without virtual planning.

All surgeries will be performed under general anesthesia using standard approaches. Clinical evaluation will include assessment of facial symmetry, eye movement, enophthalmos, diplopia, wound healing, and postoperative complications. Radiographic evaluation will be conducted by comparing postoperative 3D CT scans (after 3 months) with preoperative virtual models to assess reduction accuracy and bone formation.

Statistical Analysis:

Data will be analyzed using SPSS software. Descriptive statistics will be presented as mean ± standard deviation. Independent t-tests and ANOVA will be used to compare outcomes between groups, with significance set at p ≤ 0.05.

Expected Outcomes:

It is anticipated that virtual surgical planning will yield superior anatomical accuracy, improved facial symmetry, and reduced intraoperative time and complications compared to conventional techniques.

Ethical Approval:

Approved by the Research Ethics Committee, Faculty of Dentistry, Suez Canal University, on 30 September 2025 (Board Status: Approved).

Study Start Date: October 2025 Estimated Completion Date: October 2026

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 years) with clinically and radiographically confirmed ZMC fracture.
* Fit for general anesthesia and able to undergo CT imaging.
* Willing to sign informed consent.

Exclusion Criteria:

* Systemic diseases impairing bone healing (osteoporosis, cancer, long-term steroid use).
* Noncompliance or inability to attend follow-up visits.
* ASA class IV-VI.
* Previous facial deformities or fractures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-12-25 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Accuracy of Fracture Reduction | 3 months postoperatively
  Measurement of the 3D linear discrepancy (in millimeters) between the postoperative CT model and the preoperative virtual reduction model using surface-based 3D superimposition (color-map deviation analysis). The mean deviation (mm) will be automatically calculated by the 3D analysis software.

SECONDARY OUTCOMES:
Facial symmetry | 1 week, 1 month, and 3 months postoperatively
  Measurement of midline deviation and the distance (mm) from facial midline to the most lateral point of the malar eminence on both sides using standardized frontal photographs. Symmetry is expressed as the absolute difference in millimeters.
Eye Movement (Diplopia in Gaze Positions) | 1 week and 3 months postoperatively
  Number of the 9 standard gaze positions in which the participant reports diplopia during clinical examination. The examiner will assess ocular motility in primary position, up gaze, down gaze, right gaze, left gaze, and the 4 oblique gaze positions. Diplopia will be recorded as present or absent in each position, producing a total score from 0 to 9.
Postoperative Complications | Up to 3 months postoperatively
  Number of participants developing postoperative complications including infection, wound dehiscence, trismus, or sensory deficit. Each complication will be recorded as "yes/no" for each patient.
Surgical Time | Intraoperative (single measurement)
  Total duration of surgery recorded in minutes from initial incision to final wound closure using the operating room timing system.
Bone Healing | 3 months postoperatively
  Radiographic assessment of bone healing using postoperative CT. Bone union will be scored using a standardized 4-point CT bone healing scale (0 = no healing, 3 = complete cortical continuity).

CONTACTS AND LOCATIONS:
Overall Officials: Hossam Shaban El Fadly, principle investigator, Principal Investigator — Suez Canal University
Locations (1):
- Suez Canal University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Longeac M, Depeyre A, Pereira B, Barthelemy I, Pham Dang N. Virtual surgical planning and three-dimensional printing for the treatment of comminuted zygomaticomaxillary complex fracture. J Stomatol Oral Maxillofac Surg. 2021 Sep;122(4):386-390. doi: 10.1016/j.jormas.2020.05.009. Epub 2020 May 18. PMID 32439600
- [Result] Abdul Lateef Hassan T, Abbood Mohammed D. Virtual Surgical Planning and 3-Dimensional Printing for the Treatment of Zygomaticomaxillary Complex and/or Orbital Fracture. J Craniofac Surg. 2023 May 1;34(3):e218-e222. doi: 10.1097/SCS.0000000000009056. Epub 2022 Oct 11. PMID 36217233
- [Result] Committeri U, Magliulo R, Carraturo E, Arena A, Abbate V, Salzano G, Troise S, Barone S, Germano C, Vaira LA, Giovacchini F, Cataldo R, Grassia MG, Califano L, Piombino P. Virtual surgical planning in tripod zygomatico-maxillary complex fractures: A prospective comparison between two different strategies. J Craniomaxillofac Surg. 2024 Dec;52(12):1497-1504. doi: 10.1016/j.jcms.2024.08.020. Epub 2024 Sep 29. PMID 39349348
- [Result] Dubron K, Van Camp P, Jacobs R, Politis C, Shaheen E. Accuracy of virtual planning and intraoperative navigation in zygomaticomaxillary complex fractures: A systematic review. J Stomatol Oral Maxillofac Surg. 2022 Nov;123(6):e841-e848. doi: 10.1016/j.jormas.2022.07.003. Epub 2022 Jul 7. PMID 35809796

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form: study protocol with cover page (2025-09-30): https://cdn.clinicaltrials.gov/large-docs/33/NCT07280533/Prot_SAP_ICF_000.pdf